CLINICAL TRIAL: NCT03041506
Title: US Guided Interscalene Block Compared With Sedation for Shoulder Dislocation Reduction in the ER
Brief Title: Interscalene Nerve Block vs. Sedation for Shoulder Dislocation Reduction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TASMC-16-IM-0221-CTIL
Record Dates: First submitted 2017-01-22; First posted 2017-02-02 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Shoulder Dislocation; Brachial Plexus Block
Keywords: Shoulder dislocation reduction; Ultrasound guided interscalene block (ISCB); Sedation
MeSH Terms: conditions — Shoulder Dislocation | interventions — Lidocaine; Midazolam; Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sedation (Active Comparator): Analgesia and sedation through IV medication for pain relief will be administered to the patient.
  Midazolam: up to a maximum dosage of 0.1 mg/kg (bolus of 1 mg by titration every 30-60 second).
  Ketamine: up to maximum dosage of 100 mg IV (bolus of 25 mg by titration every 30-60 seconds).
  Interventions: Drug: Midazolam; Drug: Ketamine
- US guided ISCB (Experimental): Infiltration of local anesthetic agents around target nerves (C5, C6 nerve roots), US guidance, for shoulder pain relief and muscle relaxation.
  Lidocaine 2%: 15-20 ml.
  Interventions: Drug: Lidocaine; Procedure: US guided ISCB

INTERVENTIONS:
Drug: Lidocaine — Infiltration of local anesthetic agents around target nerves (C5, C6 nerve roots), US guidance, for shoulder pain relief and muscle relaxation.
  Lidocaine 2%: 15 -20 ml.
  Other Names: Xylocaine
  Arms: US guided ISCB
Procedure: US guided ISCB — Infiltration of local anesthetic agents around target nerves (C5, C6 nerve roots), US guidance, for shoulder pain relief and muscle relaxation.
  Lidocaine 2%: 15 -20 ml.
  Arms: US guided ISCB
Drug: Midazolam — IV administration up to a maximum dosage of 0.1 mg/kg (bolus of 1 mg by titration every 30-60 seconds) for sedation and pain relief.
  Other Names: Midolam
  Arms: Sedation
Drug: Ketamine — IV administration up to maximum dosage of 100 mg IV (bolus of 25 mg by titration every 30-60 seconds) for sedation and pain relief.
  Other Names: Ketalar
  Arms: Sedation

SUMMARY:
Shoulder dislocation is the most common joint dislocation presented to the emergency room (ER) and reduction by medical team is always needed. Shoulder dislocation and reduction are often very painful and require some form of sedation, pain relief and muscle relaxation for reduction maneuvers. Several sedation protocols for reduction maneuver are described in the literature, and each institution is guided by its own protocol to optimize patient comfort and safety. At the Tel Aviv Medical Centre (TLVMC) ER sedation with ketamine and midazolam are the mainstay form of sedation for shoulder dislocation reduction.

Sedation is not without risk, it is time consuming for the medical staff, and need personal supervision. Sedation under busy ER conditions can cause a burden to the medical team which can end up in treatment insufficiency and patient safety failure.

Ultrasound (US) guided interscalene block (ISCB) for shoulder surgery was found to be an effective method for perioperative analgesia. However, there is limited data on performance of US guided ISCB for shoulder dislocation reduction and its comparison to other analgesic modalities Both techniques (block and sedation) for shoulder dislocation procedure are being performed for two years at the TLVMC, however no study was done to evaluate these two analgesic modalities.

The current study compares sedation vs. US guided ISCB for the treatment of shoulder dislocation in the ER at the TLVMC.

Study objective:

Comparison of two common analgesic methods, Sedation vs. US guided ISCB, for shoulder dislocation reduction in our institution.

Study design:

This is a prospective, randomized, interventional, open-label study with two arms- Sedation group and US guided ISCB group. The sedation will be conducted by the orthopedic surgeon who is certified to perform sedation and the US guided ISCB will be conducted by a certified anesthesiologist.

Primary outcome:

Time frame measured from the beginning of reduction procedure until readiness for dismissal from the ER according to the physician decision.

Secondary outcomes [short list]:

Visual Analogue Score (VAS), patient satisfaction, complications, US guided ISCB and sedation failure rate, overall reduction success rate, readmission rate to the ER, daily activity level measured by Quick DASH (Disabilities of Arm, Shoulder and Hand) outcome measure.

DETAILED DESCRIPTION:
Shoulder dislocation is the most prevalent dislocation with a frequency of 0.5%-1.7% among the population, which requires reduction by medical staff in the emergency room (ER). Reduction procedure is often painful and require some level of sedation, analgesia, and muscle relaxation for its completeness. Several sedation protocols for reduction maneuver are described in the literature, and each institution is guided by its own protocol to optimize patient comfort and safety.

The literature describes multiple sedative agents such as Propofol, Etomidate, Midazolam, Fentanyl, etc. In the emergency department (ED) at Tel Aviv Medical Center (TLVMC), the sedation protocol contains Midazolam and Ketamine as the main sedative and analgesic agents.

Sedation is not without a risk. Known complications are respiratory depression, aspiration, and hemodynamic instability. These complications seem to be more prevalent in patients with decreased cardio-respiratory reserves, such as elderly, morbid obese, obstructive sleep apnea (OSA), chronic obstructive pulmonary disease (COPD) and congestive heart failure (CHF) patients.

In addition, sedation requires resources such a facility occupied with equipment for monitoring vitals, oxygen supply source, capnography and human resources including medical staff certified to provide sedation and handle any possible complication and nursing staff supervising the patient throughout the procedure from admission until release home from the ER.

The ED at the TLVMC is very active and busy throughout the day. Sedation under such condition create a real challenge for the medical team. This is translated into shortage in manpower and equipment availability and time needed to care for each patient. Such an atmosphere create huge burden on the medical team which can end up in treatment insufficiency and patient safety failure.

Recently, several new publications were published regarding the implementation of peripheral nerve block (PNB) under US guidance for analgesia and painful orthopedic procedure in the ER. Implementation of PNB for pain management in orthopedic procedures in the ER might constitute theoretical advantages over sedation.

Interscalene block (ISCB) is a very effective tool being used during shoulder surgery. However, there is limited data on performance of US guided ISCB for shoulder dislocation reduction and it's comparison with other analgesic modalities.Only one study to date compared sedation vs. US guided ISCB for shoulder dislocation reduction procedure in the ER. This study showed that patients who received ISCB had a shorter length of stay in the ER and required less supervision and medical intervention from the medical team.

Both US guided ISCB and sedation for shoulder dislocation procedure are being performed for a while at TLVMC. However no study was done to evaluate them and determine if one of the analgesic modality have any advantages over the other.

Objectives:

Comparison of two common analgesic methods, US guided ISCB vs.sedation, for shoulder dislocation reduction in the ER at the TLVMC.

Methods and Materials

Study Design:

This is a prospective, randomized, interventional non-blinded study with two arms- US guided ISCB group and Sedation group.

The sedation will be conducted by an orthopedic physician certified to perform sedation and the US guided ISCB will be conducted by an anesthesiologist who has at least one year of experience preforming regional anesthesia using US guidance.

Sample Size:

The study will include 70 subjects - 35 in each group. In order to compensate for dropouts we will aim for recruitment of 90 subjects.

Statistical Analysis:

Quantitative data with normal distribution will be evaluated using t-test for independent samples. In case the assumptions for parametric test will not hold true, quantitative data will be evaluated using an a- parametric Mann-Whitney test. Quantitative variables will be presented as mean and standard deviation.

Dichotomous data will be evaluated using chi-square test. Fischer exact test will be used when more than 20% of the expected observations were less than 5 or any expected observation was less than 2.

Categorical data will be presented as a number of cases and percent. Multivariate logistic regression analysis will be used for the primary outcome in order to determine independent risk factors. The data included in the multivariate logistic regression model will have a clinical significance according to the investigator clinical judgment and data found to have a Pv<0.1 in the univariate analysis. A Pv of 0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

1. Patients (ASA SCORE I-III) without acute cardio-pulmonary decompensation, who arrive to the ER with shoulder dislocation for reduction maneuver.

Exclusion Criteria:

1. Unconscious patient
2. Patient refusal/unable to give informed consent
3. Patients with acute cardio-pulmonary decompensation
4. Patients with known allergy to medications which will be included in the study
5. Patients who suffer additional injuries and need to be hospitalized for further treatment
6. Patients who received narcotic/sedative premedication before the procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-02-15 (Estimated); Primary Completion 2017-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Length of stay measured in minutes from the beginning of shoulder dislocation reduction procedure until the subject is ready for discharge from the ER according to the physician decision | Up to 3 hours from shoulder dislocation reduction procedure

SECONDARY OUTCOMES:
Visual Analogue Score (VAS) before the shoulder dislocation reduction procedure | Baseline
Visual Analogue Score (VAS) when subject is ready for discharge from the ER according to the physician decision | When subject is ready for discharge from the ER according to the physician decision, up to 3 hours from shoulder dislocation reduction procedure
Patient satisfaction from shoulder dislocation reduction procedure when subject is ready for discharge from the ER according to the physician decision | When subject is ready for discharge from the ER according to the physician decision, up to 3 hours from shoulder dislocation reduction procedure
Side effect and complications related to US guided ISCB during shoulder dislocation reduction procedure | During shoulder dislocation reduction procedure
  1. Pneumothorax - clinical symptoms of dyspnea, hypoxemia, tachypnea + radiologic confirmation of pneumothorax
  2. Local anesthetic systemic toxicity - clinical symptoms range from tinnitus, metallic taste, seizures, loss of consciousness, cardiac arrhythmias, and cardiac arrest
  3. Intrathecal injection - local anesthetics penetrate into the subarachnoid space resulting in high spinal anesthesia
  4. Intravascular puncture - blood appear in the syringe
  5. Horner syndrome - ptosis, miosis and anhydrosis ipsilateral to the side of the ISCB
  6. Hoarseness - voice change
  7. Respiratory failure - phrenic nerve blockade with resultant diaphragmatic paresis in the ipsilateral side of the ISCB
  8. Neurologic injury - sensory or motor deficit after ISCB
Complications related to sedation during shoulder dislocation reduction procedure | During shoulder dislocation reduction procedure
  1. Respiratory complications - aspiration with signs of fluid or food regurgitation respiratory depression and upper airway obstruction
  2. Hemodynamic instability - cardiac arrhythmias and hypotension
Failed US guided ISCB rate (preceded by sedation) during shoulder dislocation reduction procedure | During shoulder dislocation reduction procedure
  Failed ISCB - no loss of cold sensation over the blocked shoulder and no pain relief after ISCB
Overall success rate for shoulder dislocation reduction procedure | During shoulder dislocation reduction procedure
  Success full shoulder reduction - confirmed by an X ray study
Easiness of shoulder dislocation reduction procedure assessed by orthopedic physician | During shoulder dislocation reduction procedure
  The orthopedic physician will be asked to describe his/her personal difficulty to perform the shoulder dislocation reduction procedure Severity score: 1-Easy; 2-Relatively easy; 3-Moderate; 4-Moderate to severe; 5-Severe
Failed sedation rate (preceded by general anesthesia) during shoulder dislocation reduction procedure | During shoulder dislocation reduction procedure
  Failed sedation - patient is uncooperative or in pain not allowing the orthopedic physician to perform reduction procedure
Visual Analogue Score (VAS) 24 hours after readiness for dismissal from ER | 24 hours after readiness for dismissal
Readmission to the ER during 24 hours from readiness for dismissal from the ER | During 24 hours from readiness for dismissal
  Any reason for patient readmission to the ER
Limb daily activity level measured by "Quick DASH" score 72 hours from readiness for dismissal from the ER | 72 hours from readiness for dismissal from the ER
  Quick DASH is a questionnaire that measure upper limb daily activity level

CONTACTS AND LOCATIONS:
Overall Officials: Idit Matot, MD, Principal Investigator — Chair, Division of Anesthesiology & Critical Care & Pain Tel-Aviv Sourasky Medical Center

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual participant data (IPD).

REFERENCES:
- [Background] Perron AD, Ingerski MS, Brady WJ, Erling BF, Ullman EA. Acute complications associated with shoulder dislocation at an academic Emergency Department. J Emerg Med. 2003 Feb;24(2):141-5. doi: 10.1016/s0736-4679(02)00717-5. PMID 12609642
- [Background] Orlinsky M, Shon S, Chiang C, Chan L, Carter P. Comparative study of intra-articular lidocaine and intravenous meperidine/diazepam for shoulder dislocations. J Emerg Med. 2002 Apr;22(3):241-5. doi: 10.1016/s0736-4679(01)00475-9. PMID 11932085
- [Background] Matthews DE, Roberts T. Intraarticular lidocaine versus intravenous analgesic for reduction of acute anterior shoulder dislocations. A prospective randomized study. Am J Sports Med. 1995 Jan-Feb;23(1):54-8. doi: 10.1177/036354659502300109. PMID 7726351
- [Background] Burton JH, Bock AJ, Strout TD, Marcolini EG. Etomidate and midazolam for reduction of anterior shoulder dislocation: a randomized, controlled trial. Ann Emerg Med. 2002 Nov;40(5):496-504. doi: 10.1067/mem.2002.126607. PMID 12399793
- [Background] Taylor DM, O'Brien D, Ritchie P, Pasco J, Cameron PA. Propofol versus midazolam/fentanyl for reduction of anterior shoulder dislocation. Acad Emerg Med. 2005 Jan;12(1):13-9. doi: 10.1197/j.aem.2004.08.039. PMID 15635132
- [Background] Roback MG, Wathen JE, Bajaj L, Bothner JP. Adverse events associated with procedural sedation and analgesia in a pediatric emergency department: a comparison of common parenteral drugs. Acad Emerg Med. 2005 Jun;12(6):508-13. doi: 10.1197/j.aem.2004.12.009. PMID 15930401
- [Background] Blaivas M, Lyon M. Ultrasound-guided interscalene block for shoulder dislocation reduction in the ED. Am J Emerg Med. 2006 May;24(3):293-6. doi: 10.1016/j.ajem.2005.10.004. PMID 16635700
- [Background] Beaudoin FL, Nagdev A, Merchant RC, Becker BM. Ultrasound-guided femoral nerve blocks in elderly patients with hip fractures. Am J Emerg Med. 2010 Jan;28(1):76-81. doi: 10.1016/j.ajem.2008.09.015. PMID 20006206
- [Background] Reid N, Stella J, Ryan M, Ragg M. Use of ultrasound to facilitate accurate femoral nerve block in the emergency department. Emerg Med Australas. 2009 Apr;21(2):124-30. doi: 10.1111/j.1742-6723.2009.01163.x. PMID 19422409
- [Background] Abrahams MS, Aziz MF, Fu RF, Horn JL. Ultrasound guidance compared with electrical neurostimulation for peripheral nerve block: a systematic review and meta-analysis of randomized controlled trials. Br J Anaesth. 2009 Mar;102(3):408-17. doi: 10.1093/bja/aen384. Epub 2009 Jan 26. PMID 19174373
- [Background] Neal JM, Barrington MJ, Brull R, Hadzic A, Hebl JR, Horlocker TT, Huntoon MA, Kopp SL, Rathmell JP, Watson JC. The Second ASRA Practice Advisory on Neurologic Complications Associated With Regional Anesthesia and Pain Medicine: Executive Summary 2015. Reg Anesth Pain Med. 2015 Sep-Oct;40(5):401-30. doi: 10.1097/AAP.0000000000000286. PMID 26288034
- [Background] Borgeat A, Ekatodramis G. Anaesthesia for shoulder surgery. Best Pract Res Clin Anaesthesiol. 2002 Jun;16(2):211-25. doi: 10.1053/bean.2002.0234. PMID 12491553
- [Background] Singelyn FJ, Lhotel L, Fabre B. Pain relief after arthroscopic shoulder surgery: a comparison of intraarticular analgesia, suprascapular nerve block, and interscalene brachial plexus block. Anesth Analg. 2004 Aug;99(2):589-92, table of contents. doi: 10.1213/01.ANE.0000125112.83117.49. PMID 15271745
- [Background] Davis JJ, Swenson JD, Greis PE, Burks RT, Tashjian RZ. Interscalene block for postoperative analgesia using only ultrasound guidance: the outcome in 200 patients. J Clin Anesth. 2009 Jun;21(4):272-7. doi: 10.1016/j.jclinane.2008.08.022. Epub 2009 Jun 6. PMID 19502031
- [Background] Liu SS, Zayas VM, Gordon MA, Beathe JC, Maalouf DB, Paroli L, Liguori GA, Ortiz J, Buschiazzo V, Ngeow J, Shetty T, Ya Deau JT. A prospective, randomized, controlled trial comparing ultrasound versus nerve stimulator guidance for interscalene block for ambulatory shoulder surgery for postoperative neurological symptoms. Anesth Analg. 2009 Jul;109(1):265-71. doi: 10.1213/ane.0b013e3181a3272c. PMID 19535720
- [Background] Blaivas M, Adhikari S, Lander L. A prospective comparison of procedural sedation and ultrasound-guided interscalene nerve block for shoulder reduction in the emergency department. Acad Emerg Med. 2011 Sep;18(9):922-7. doi: 10.1111/j.1553-2712.2011.01140.x. Epub 2011 Aug 30. PMID 21883635